CLINICAL TRIAL: NCT04054596
Title: Strategy Based Technique to Enhance Memory (STEM) for Improving New Learning and Memory (NLM) in Moderate to Severe TBI: A Randomized Clinical Trial
Brief Title: Strategy Based Technique to Enhance Memory (STEM) for Improving New Learning and Memory (NLM) in Moderate to Severe TBI
Acronym: STEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nancy Chiaravalloti, Director of NNL & TBI, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-993-17
Record Dates: First submitted 2019-06-18; First posted 2019-08-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injury; Cognitive Impairment
Keywords: Traumatic Brain Injury; Cognitive Impairment; Intervention
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The purpose of this research study is to investigate the effectiveness of a memory enhancement technique in persons with a Traumatic Brian Injury (TBI).
Who Masked: Participant, Outcomes Assessor
Masking Description: Once enrolled, participants will be randomly assigned to the TX or CTL group via a computerized random number generator coordinated by the statistician, who will not be blinded. Group assignment will be concealed. Both the participant and the examiner conducting the baseline and outcome assessments will be blind to group membership.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STEM (Experimental): The treatment group (TX) will complete 8 sessions of STEM (2 sessions per week for 4 weeks), Sessions are approximately 30-45 minutes long.
  Interventions: Behavioral: SME
- Controlled (No Intervention): During weeks 2-5, one group will undergo a memory enhancement protocol, used to improve memory functioning in individuals with neurological injuries. The other group will serve as a control group and complete memory exercises with the researcher.

INTERVENTIONS:
Behavioral: SME — The treatment group (TX) will complete 8 sessions of SME (2 sessions per week for 4 weeks), de-signed to teach the concepts of SG, SL and RP and the application of these techniques in daily life. Sessions are approximately 30-45 minutes long.
  Arms: STEM

SUMMARY:
The purpose of this research study is to investigate the effectiveness of a memory enhancement technique in persons with a Traumatic Brian Injury (TBI). The study is designed to research how well this technique can help people with TBI improve their memory and their ability to function better in everyday life

DETAILED DESCRIPTION:
Impairments in higher level cognitive processing, such as new learning and memory, are common in Traumatic Brain Injury (TBI)and negatively impact multiple aspects of everyday life, including occupational and social functioning. Despite this, few studies have attempted to remediate these cognitive deficits in order to improve everyday functioning. While not applied in traditional rehabilitation protocols as of yet, many techniques from cognitive psychology significantly improve learning and memory in healthy persons. These techniques include the generation effect (GE), the spacing effect (SE), and the testing effect (TE). These techniques have recently been incorporated into an 8-session treatment protocol, Stylistic Memory Enhancement (SME), designed to teach participants about each of the techniques, train them on how to apply the techniques in daily life and practice their application to daily life memory demanding situations. The protocol includes teaching participants how to restructure a memory demanding situation in order to make optimal use of self-generation, spaced learning and self-testing.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study I must meet the following requirements:

* I am between the ages of 18-65.
* I have had a traumatic brain injury (TBI) at least 1 year ago.
* I can read and speak English fluently.
* I have difficulties with learning and memory skills.

Exclusion Criteria:

* I have had a prior stroke or neurological injury/disease other than TBI.
* I have a history of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder, Schizophrenia, Bipolar Disorder I or II.
* I have a significant alcohol or drug abuse history (inpatient Treatment).
* I am taking certain medications that might exclude me from the research. The study team will review my medications with me.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Self Report Deficits in Daily Life | 5 weeks from baseline (short term follow-up) and 7 months from baseline (long term follow-up)
  Perceived Deficits Questionnaire215
  * •20 items; evaluates everyday situations in which cognition has a role
  * •Cronbach's Alpha (lower bound reliability) = .93

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Chiaravalloti, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States